CLINICAL TRIAL: NCT01548742
Title: Meditation Interventions for Treatment of PTSD in Veterans
Acronym: VMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPLE-012-11S; CX-11-012 (Other Grant/Funding Number: VA Clinical Science Research & Development (CSR&D))
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Meditation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Mindfulness-Based Stress Reduction (MBSR) (Experimental): Mindfulness-Based Stress Reduction (MBSR)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Arm 2: Present-Centered Group Therapy (PCGT) (Active Comparator): Present-Centered Group Therapy (PCGT)
  Interventions: Behavioral: Present-Centered Group Therapy (PCGT)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Mindfulness Based Stress Reduction (MBSR) is a group based treatment focused on progressive training in mindfulness meditation.
  Other Names: MBSR
  Arms: Arm 1: Mindfulness-Based Stress Reduction (MBSR)
Behavioral: Present-Centered Group Therapy (PCGT) — Present-Centered Group Therapy (PCGT) is a group therapy focused on current problems.
  Arms: Arm 2: Present-Centered Group Therapy (PCGT)

SUMMARY:
Posttraumatic stress disorder (PTSD) is a debilitating psychiatric disorder which results in serious impairments in interpersonal, occupational and social functioning. Effective treatments are available for PTSD but they do not work for everyone. Alternative treatments are needed to help those veterans not helped by currently available treatments. Mindfulness Based Stress Reduction (MBSR) is a group based treatment focused on mindfulness meditation. MBSR has been found to be effective in helping people with problems with pain and anxiety. MBSR has not yet been studied in veterans with PTSD. The proposed study will compare MBSR with a standard psychotherapy treatment in veterans with PTSD. This research is relevant to Veterans' health because of the need to develop alternative treatments for veterans with PTSD who have not responded to currently available treatments.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a debilitating psychiatric disorder associated with high rates of chronicity, poor quality of life, and severe impairments in interpersonal, occupational, and social functioning. While evidence-based psychotherapies for treatment of PTSD have been developed and disseminated within the VA system, no treatment has shown universal effectiveness and there have been great concerns about attenuated treatment response and elevated treatment drop out in veteran populations. The evaluation of alternative treatment modalities for veterans with PTSD is therefore an important priority. The Minneapolis VA Health Care System (MVAHCS) has taught Mindfulness Based Stress Reduction (MBSR), a group-based intervention focused on mindfulness meditation, to veteran clinical populations since 2001, and pilot data from veterans diagnosed with PTSD is promising. Despite support for the application of MBSR to other mental health and physical problems, MBSR has not been systematically evaluated as a treatment for PTSD. Moreover, the existing literature on MBSR is limited by methodological weaknesses. If shown to be efficacious through scientifically sound trials, MSBR may offer an effective, acceptable, and tolerable intervention for veterans suffering PTSD who are unable to engage in or complete traditional exposure-based therapies. The primary goal of this proposal is to conduct a methodologically rigorous randomized controlled trial (RCT) of MBSR in treating PTSD among veterans, examining both symptom outcomes and subsequent health services utilization. Given our compelling pilot data, we propose initial steps to evaluate putative mechanisms of change (self-report and electrophysiology markers, i.e., EEG) through which MBSR may relate to PTSD symptom improvements, and to examine the acceptability of MBSR to the veteran population.

The MVAHCS and the assembled team combines expertise in PTSD treatment and research, clinical trials, and neuroscience, with clinical expertise in MBSR and compelling pilot data to support the feasibility and scope of the current project. The efficacy of MBSR will be examined relative to present-centered group therapy (PCGT), a non-specific therapeutic comparison group. Veterans diagnosed with PTSD will be randomized to MBSR or PCGT for 9 weeks. Each intervention will be delivered in group format following manualization by trained clinicians receiving expert supervision. Treatment integrity will be independently monitored. Assessment of clinical outcomes post-treatment and 2 months follow-up will be independently evaluated. Putative mechanisms of mindfulness meditation will be assessed using self-report and electrophysiology markers. We have the following aims:

Primary Aim 1: To evaluate the efficacy of MBSR as a treatment for PTSD in veterans compared to PCGT over 9-weeks of treatment and 2-month follow-up.

Secondary Aim 1: To identify potential treatment-based predictors of PTSD outcomes.

Secondary Aim 2: To identify differences in subsequent VA health services utilization among veterans across treatment conditions.

Exploratory Aims:

1. To evaluate rates of drop-out, compliance, and consumer satisfaction with MBSR.
2. To evaluate acceptability and outcomes of treatment with veterans with mild traumatic brain injuries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female veterans who are 18 years or older.
* Must meet current DSM-IV criteria for PTSD based on the Clinician Administered PTSD Scale (CAPS) or have a PTSD Checklist (PCL) score between 40 and 60.
* If taking psychoactive medications, must be on a stable regime for 8 weeks or more.

Exclusion Criteria:

* Current suicidal or homicidal ideation with intent and/or plan that, in the judgment of the investigator, should be the focus of treatment.
* Current substance dependence (not in sustained remission), current or recent (within past 6 months) manic episode, or active psychosis. To be eligible, if veteran has current diagnosis of bipolar disorder, there is evidence that illness has been stable for at least 6 months on medication. Has unstable or serious medical illness, including history of stroke, seizure disorder, or unstable cardiac disease that would interfere with participation in treatment.
* Severe cognitive impairment or moderate/severe traumatic brain injury.
* Unable to comprehend or communicate in English.
* Unwilling to accept random assignment or unwilling to refrain from participating in other active forms of psychotherapy during 8-week treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- VA Medical Center, Minneapolis, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Shapira I, Richman J, Pace TWW, Lim KO, Polusny MA, Hamner MB, Bremner JD, Mumba MN, Jacobs ML, Pilkinton P, Davis LL. Biomarker Response to Mindfulness Intervention in Veterans Diagnosed with Post-traumatic Stress Disorder. Mindfulness (N Y). 2022 Oct;13(10):2448-2460. doi: 10.1007/s12671-022-01969-6. Epub 2022 Sep 12. PMID 36938380
- [Derived] Kang SS, Sponheim SR, Lim KO. Interoception Underlies Therapeutic Effects of Mindfulness Meditation for Posttraumatic Stress Disorder: A Randomized Clinical Trial. Biol Psychiatry Cogn Neurosci Neuroimaging. 2022 Aug;7(8):793-804. doi: 10.1016/j.bpsc.2021.10.005. Epub 2021 Oct 21. PMID 34688923
- [Derived] Polusny MA, Erbes CR, Thuras P, Moran A, Lamberty GJ, Collins RC, Rodman JL, Lim KO. Mindfulness-Based Stress Reduction for Posttraumatic Stress Disorder Among Veterans: A Randomized Clinical Trial. JAMA. 2015 Aug 4;314(5):456-65. doi: 10.1001/jama.2015.8361. PMID 26241597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through flyers posted in targeted clinics and clinical referrals at the Minneapolis VA Medical Center.
Pre-assignment Details: Participants completed a 5-hour eligibility and baseline assessment that included a structured clinical interview and self-report measures. Randomization occurred for those meeting study inclusion criteria.
Period: Overall Study
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT)
Started | 58 | 58
Completed | 45 | 54
Not Completed | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT) | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.4) | 59.4 (9.2) | 58.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 46 | 52 | 98
Race/Ethnicity, Customized [Number; unit: participants]
  White | 47 | 50 | 97
  Black | 3 | 6 | 9
  Other | 2 | 2 | 4
  Mixed | 6 | 0 | 6
Service Era [Number; unit: participants]
  OEF/OIF | 6 | 5 | 11
  Gulf War | 9 | 8 | 17
  Vietnam War | 41 | 45 | 86
  Other | 2 | 0 | 2
Lifetime trauma exposure [Mean (Standard Deviation); unit: No. of events] | 7.9 (3.3) | 7.5 (3.0) | 7.7 (3.1)
Lifetime trauma exposure event type [Number; unit: participants]
  Combat exposure | 39 | 47 | 86
  Sexual trauma | 21 | 11 | 32
  Physical assault | 39 | 37 | 76
  Disaster exposure | 25 | 25 | 50
  Serious accident | 38 | 36 | 74
  Life-threatening illness or injury | 34 | 33 | 67
  Other traumatic event | 55 | 55 | 110
PTSD diagnosis [Number; unit: participants] — Full PTSD criteria defined according to the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) (DSM-IV). Subthreshold PTSD defined as endorsement of DSM-IV criterion A1 and at least 1 symptom each from criteria B, C, and D with significant impairment.
  participants
    Full PTSD criteria | 57 | 56 | 113
    Subthreshold PTSD | 1 | 2 | 3
Comorbid mood disorder [Number; unit: participants] | 26 | 23 | 49
Taking psychotropic medication [Number; unit: participants] | 51 | 49 | 100
Total number of psychotherapy mental health visits [Mean (Standard Deviation); unit: sessions] | 13.2 (28.3) | 14.6 (29.2) | 13.9 (28.7)
Duration of previous mental health care [Mean (Standard Deviation); unit: months] | 69.0 (53.3) | 63.9 (45.2) | 66.5 (9.2)
Number of participants receiving 8 or more therapy sessions in PTSD or mental health clinics [Number; unit: participants] | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms on the PTSD Checklist (PCL) at Baseline, During Treatment, After Treatment and at 2-Month Follow-up
Description: The PCL is a valid and reliable measure of PTSD symptoms. Score range from 17-85; higher scores indicate more severe symptoms. The minimal clinically important difference for self-reported PTSD symptom severity is a reduction of 10 or more points on the PCL.
Time Frame: Baseline, Weeks 3, 6, 9 and 17
Population: Intent to treat population (all participants randomized to treatment).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT)
Number analyzed (Participants) | 58 | 58
units on a scale
  Baseline PCL | 63.6 [60.6 to 66.7] | 58.8 [55.7 to 61.8]
  Week 3 PCL | 63.9 [60.8 to 67.0] | 61.7 [58.6 to 64.8]
  Wee 6 PCL | 61.3 [58.1 to 64.4] | 60.7 [57.6 to 63.8]
  Week 9 PCL | 55.7 [52.6 to 58.9] | 55.8 [52.7 to 58.9]
  Week 17 PCL | 54.4 [51.2 to 57.6] | 56.0 [52.9 to 59]

2. Other Pre Specified Outcome: Clinically Significant Improvement in Self-reported PTSD Symptoms as Measured by the PCL
Description: % of participants with clinically significant improvement in self-reported PTSD symptoms defined as a reduction of 10 points or more on the PCL.
Time Frame: Weeks 9 and 17
Population: Intent to treat analysis
Measure: Number (95% Confidence Interval); unit: percentage clinical responders
Groups:
- Arm 1: Mindfulness Based Stress Reduction (MBSR): Mindfulness-Based Stress Reduction (MBSR): Mindfulness Based Stress Reduction (MBSR) is a group based treatment focused on progressive training in mindfulness meditation.
- Arm 2: Present Centered Group Therapy (PCGT): Present-Centered Group Therapy (PCGT): Present-Centered Group Therapy (PCGT) is a group therapy focused on current problems.
Arm/Group | Arm 1: Mindfulness Based Stress Reduction (MBSR) | Arm 2: Present Centered Group Therapy (PCGT)
Number analyzed (Participants) | 58 | 58
percentage clinical responders
  % responders, Week 9 | 36.5 [24 to 49] | 22.8 [10.9 to 34.7]
  % responders, Week 17 | 48.9 [35.1 to 62.8] | 28.1 [15.5 to 40.6]

3. Secondary Outcome: PTSD Symptom Severity on the Clinician Administered PTSD Scale (CAPS) at Baseline, After Treatment, and at 2-Month Follow-up
Description: The CAPS is a valid and reliable measure of PTSD symptom severity. Score range from 0-136; higher scores indicate more severe symptoms. The minimal clinically important difference for self-reported PTSD symptom severity is a reduction of 10 or more points on the CAPS.
Time Frame: Baseline, Weeks 9 and 17
Population: Intent to treat population (all participants randomized to treatment).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT)
Number analyzed (Participants) | 58 | 58
units on a scale
  Baseline CAPS | 69.9 [65.0 to 74.8] | 62.5 [57.6 to 67.4]
  Week 9 CAPS | 56.3 [51.0 to 61.5] | 51.7 [46.5 to 56.8]
  Week 17 CAPS | 49.8 [44.3 to 55.3] | 50.6 [45.4 to 55.8]

4. Secondary Outcome: Depression Symptom Severity on the Patient Health Questionnaire-9 (PHQ-9) at Baseline, After Treatment, and at 2-Month Follow-up
Description: The PHQ-9 is a valid and reliable measure of depression symptom severity. Score range from 0-27; higher scores indicate more severe symptoms. The minimal clinically important difference for self-reported PTSD symptom severity is a reduction of 5 or more points on the PHQ-9.
Time Frame: Baseline, Weeks 9 and 17
Population: Intent to treat population (all participants randomized to treatment).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT)
Number analyzed (Participants) | 58 | 58
units on a scale
  Baseline PHQ-9 | 15.5 [13.9 to 17.0] | 14.6 [13.1 to 16.2]
  Week 9 PHQ-9 | 13.6 [12.0 to 15.1] | 13.9 [12.3 to 15.4]
  Week 17 PHQ-9 | 13.3 [11.7 to 15.0] | 13.8 [12.2 to 15.4]

5. Other Pre Specified Outcome: Clinically Significant Improvement in Clinician Administered PTSD Scale (CAPS)
Description: % of participants with clinically significant improvement in interviewer-rated PTSD symptom severity defined as a reduction of 10 points or more on the CAPS.
Time Frame: Weeks 9 and 17
Population: Intent to treat analysis
Measure: Number (95% Confidence Interval); unit: percentage clinical responders
Arm/Group | Arm 1: Mindfulness Based Stress Reduction (MBSR) | Arm 2: Present Centered Group Therapy (PCGT)
Number analyzed (Participants) | 58 | 58
percentage clinical responders
  % responders, Week 9 | 63.5 [49.8 to 77.1] | 49.1 [36.1 to 62.1]
  % responders, Week 17 | 66.7 [52.1 to 81.2] | 54.5 [41.4 to 67.7]

ADVERSE EVENTS:
Arm/Group | Arm 1: Mindfulness-Based Stress Reduction (MBSR) | Arm 2: Present-Centered Group Therapy (PCGT)
Serious Adverse Events (participants affected / at risk) | 1/58 | 2/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Mindfulness-Based Stress Reduction (MBSR) (N=58) | Arm 2: Present-Centered Group Therapy (PCGT) (N=58)
Suicide Attempt or worsening of symptoms (Psychiatric disorders) | 1 (1) | 1 (1) — Resulted in inpatient hospitalization.
Crushed by falling tree (General disorders) | 0 | 1 (1) — Survived with multiple physical injuries

LIMITATIONS AND CAVEATS:
Initial analyses did not account for clustering effects. However, when we re-analyzed data using a multilevel model including a random effect for therapy group, we found that the results were essentially unchanged.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No